CLINICAL TRIAL: NCT00686452
Title: Airway Dysfunction and Remodelling in Athletes Following Swimming Training in Chlorinated Pools
Acronym: proto nage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Dr Louis-Philippe BOULET, MD, Hôpital Laval
Other Study IDs: CER20159
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-05

CONDITIONS: Asthma; Airway Hyperresponsiveness
Keywords: Asthma; Airway hyperresponsiveness; Swimmers; Airway inflammation; Airway remodelling
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity; Airway Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, bronchial biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 1: Swimmers without AHR
- 2: Swimmers with asymptomatic AHR
- 3: Swimmers with symptomatic AHR and use only of beta-2 adrenargic
- 4: Swimmers with asthma and inhaled corticosteroids
- 5: Healthy Subjects
- 6: Healthy subjects with AHR
- 7: Healthy subjects with symptomatic AHR (asthma) but without treatment

SUMMARY:
Swimmers show the highest prevalence of asthma among elite athletes, certainly due to chlorine exposure. The consequences of a chronic exposure to chlorine compounds by swimmers and the mechanisms of asthme in this population are still poorly documented. Specific diagnostic criteria have been proposed by the International Olympic Committee - Medical Council (IOC-MC) and World anti-doping agency (WADA) to determine the presence of asthma in athletes. Using the more specific bronchial provocation tests, our aims are

1. to compare the prevalence of asthma in swimmers and control subjects
2. to analyze the Influence of chlorine exposure on bronchial inflammatory processes in swimmers versus control subjects
3. to study the time-course of changes in airway symptoms, responsiveness, inflammation and remodeling after cessation of training

ELIGIBILITY:
Inclusion Criteria:

* 14 to 35 years old
* To swim at least 10h per week
* For control subjects, non-competitive healthy subjects

Exclusion Criteria:

* any disease that may interfere with the tests for the controls
* Triathletes are excluded
* Smokers
* Obese or with a BMI more than 29
* Former athletes (control group)

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Swimmers from Quebec swimming school and universities Control from université Laval or secondary School
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Asthma and airway hyperreactivity prevalence in swimmers | 3 measurements in the year

SECONDARY OUTCOMES:
Airway inflammation and remodeling in swimmers | 3 measurements in the year and a bronchial biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche en pneumologie et en cardiologie de l'hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Bougault V, Odashiro P, Turmel J, Orain M, Laviolette M, Joubert P, Boulet LP. Changes in airway inflammation and remodelling in swimmers after quitting sport competition. Clin Exp Allergy. 2018 Dec;48(12):1748-1751. doi: 10.1111/cea.13257. Epub 2018 Sep 14. No abstract available. PMID 30141830
- [Derived] Bougault V, Turmel J, Boulet LP. Bronchial challenges and respiratory symptoms in elite swimmers and winter sport athletes: Airway hyperresponsiveness in asthma: its measurement and clinical significance. Chest. 2010 Aug;138(2 Suppl):31S-37S. doi: 10.1378/chest.09-1689. Epub 2010 Apr 2. PMID 20363843